CLINICAL TRIAL: NCT04328246
Title: The PROTECT Study: Pressure injuRy preventiOn by inTermittent EleCtrical sTimulation
Brief Title: Pressure injuRy preventiOn by inTermittent EleCtrical sTimulation
Acronym: PROTECT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment was not feasible at site.
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Rehabtronics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0018
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2020-03

CONDITIONS: Pressure Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IES Device + Standard of Care (Experimental): Intermittent electrical stimulation system. Charged pulses will be administered to bilateral gluteus maximus through surface electrodes. Stimulation occurs at 30 Hz for 10s every 10 minutes. The intervention is administered 24/7 and added to the standard of care management. Standard of care is defined as turning the patient every two hours.
  Interventions: Device: IES System; Other: Standard of Care Therapy
- Standard of Care (Active Comparator): Standard of care treatment for pressure injuries is turning the patient every two hours.
  Interventions: Other: Standard of Care Therapy

INTERVENTIONS:
Device: IES System — The IES system is composed of a stimulator and self-adhesive surface gel electrodes.
  Arms: IES Device + Standard of Care
Other: Standard of Care Therapy — Standard institutional practices for treating pressure injury.

SUMMARY:
The proposed study assesses the superiority of IES supplementation to the standard of care alone (offloading pressure every two hours) in improving the prevention and treatment of sacral and ischial pressure injuries.

ELIGIBILITY:
Inclusion Criteria:

1. Modified Braden Scale score of 14 or less. The Modified Braden Scale score is calculated as follows:

   Braden Scale score (Ranges from 6 to 23)
   * 1 for Low Serum Albumin
   * 1 for Type II Diabetes
2. Anticipated length of stay of at least 4 days
3. BMI < 35
4. Participants capable of giving informed consent, or if appropriate, participants having an acceptable individual capable of giving consent on the participant's behalf.

Exclusion Criteria:

1. Existing pressure injuries above Stage II and injuries classified as DTI or unstageable
2. Neuromuscular blocking drugs & myasthenia gravis: may prevent the ability of electrical stimulation to induce muscular contraction
3. Unstable spinal, pelvic, or hip fractures that may be displaced by a forced contraction
4. Rhabdomyolysis
5. Use of a Pacemaker
6. Skin breakdown over the gluteal regions that would preclude the use of surface electrodes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Clinical course of pressure injury over time | Patients will be assessed daily for pressure injury location and stage through treatment completion, an average of 14 days.
  Chauhan Weighted Trajectory Analysis (CWTA) will be used to compare the morbidity associated with sacral and ischial pressure injuries through time. A one-sided Chauhan logrank test at a significance of 0.05 will be used to assess for superiority of the experimental arm over the control arm.

SECONDARY OUTCOMES:
Clinical course of pressure injury in subgroups | Patients will be assessed daily for pressure injury location and stage through treatment completion, an average of 14 days.
  Chauhan Weighted Trajectory Analysis (CWTA) will be used to compare the morbidity associated with sacral and ischial pressure injuries through time. A one-sided Chauhan logrank test at a significance of 0.05 will be used to assess superiority.
Kaplan-Meier Time-to-Event Analysis | Final analysis will be performed at end of study (expected completion 2 years)
  A Kaplan Meier Curve and logrank Test (one-sided significance at p < 0.05) will be used to evaluate a difference in sacral and ischial pressure injury time-to-event morbidity between groups. An "event" is defined as the development of any stage/class of pressure ulcer.
Cox Regression Analysis | Final analysis will be performed at end of study (expected completion 2 years)
  Cox-regression analysis will be used to determine whether the implementation of the IES device is associated with a significant difference in sacral and ischial pressure injury time-to-event occurrence between treatment groups.
Observed Counts of Pressure Injuries | Final analysis will be performed at end of study (expected completion 2 years)
  Descriptive statistics and Chi-square testing will be used to compare in incidence rates and proportion between the treatment groups for sacral and ischial pressure injuries classified as Stage I-IV or Unstageable
Onset Time | Final analysis will be performed at end of study (expected completion 2 years)
  Descriptive statistics will be used to report the central tendency and spread of the onset time of a sacral and ischial pressure injury for both treatment groups and for injuries classified as Stage I-IV or Unstageable
Relative Risk | Final analysis will be performed at end of study (expected completion 2 years)
  Relative risk of sacral and ischial pressure injuries will be compared between treatment groups using a 2x2 contingency table with a 95% confidence interval.
Duration of Inpatient Stay | Final analysis will be performed at end of study (expected completion 2 years)
  Descriptive statistics will be used to report the central tendency and spread of the duration of inpatient stay for both treatment groups
Description of adverse events related to IES | Final analysis will be performed at end of study (expected completion 2 years)
  We will report frequency and severity of skin changes underlying the electrodes, categorized as i) transient erythema after electrode removal, ii) non-transient skin changes after electrode removal, iii) skin breakdown under electrode.

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada